CLINICAL TRIAL: NCT02320799
Title: Randomized Controlled Trial of Interpersonal Psychotherapy for Depression and PTSD Among HIV-infected Women Exposed to Gender Based Violence in Kenya
Brief Title: Randomized Controlled Trial of Interpersonal Psychotherapy for Depression and PTSD Among HIV+ Women in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23MH098767-01A1 (NIH); K23MH098767 (NIH)
Record Dates: First submitted 2014-09-09; First posted 2014-12-19 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Depression; Posttraumatic Stress Disorder; HIV
Keywords: interpersonal psychotherapy; HIV; women; gender based violence; mental health; africa; kenya; global mental health; HIV treatment adherence
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Psychological Well-Being | interventions — Interpersonal Psychotherapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment as usual (Active Comparator): Usual Clinic psychosocial treatment
  Interventions: Behavioral: treatment as usual
- interpersonal psychotherapy (Experimental): Interpersonal Psychotherapy is an evidence-based structured, brief psychotherapy which focuses on improving relationships in order to improve mood and reduce anxiety.
  Interventions: Behavioral: interpersonal psychotherapy

INTERVENTIONS:
Behavioral: interpersonal psychotherapy — Interpersonal psychotherapy is an evidence based, structured, brief psychotherapy which improves relationships in order to improve mood and reduce anxiety
  Arms: interpersonal psychotherapy
Behavioral: treatment as usual — Clinic psychosocial treatment as usual
  Arms: treatment as usual

SUMMARY:
The aim of this study is to conduct a 12-week IPT+TAU versus wait list TAU in a cohort of HIV+GBV+ women in Nyanza Province to relieve depression and PTSD and improve ARV adherence. This pilot study will provide data on the efficacy trends, acceptability and feasibility of our IPT intervention and will generate preliminary findings for an R01-funded intervention to test the intervention's efficacy for remediating the effects of GBV trauma on mental health and HIV-related outcomes.

Hypothesis 1: IPT+ TAU will be more effective for reduction of depression and PTSD than TAU alone.

Hypothesis 2: IPT+TAU will be acceptable and feasible.

DETAILED DESCRIPTION:
We will use a parallel design with FACES Treatment as Usual (TAU) control to provide IPT once per week for twelve weeks to HIV+GBV+ women meeting CIDI diagnostic criteria for depression (MDD, dysthymia, minor depression) and PTSD secondary to GBV. Blocked randomization will be used to evenly distribute 120 participants to (1) IPT + TAU or (2) TAU for 12 weeks. The TAU group will be offered IPT treatment following the initial 12 week trial. Thus, all study subjects will receive TAU throughout the study and they will all receive IPT in either the first or second half of the study. My research team at FACES will be recruited for IPT training as potential therapists in the IPT pilot. A run-in study design will be used, assigning one training case apiece to each of the 8 therapists to practice IPT skills. Both IPT + TAU and TAU groups will be measured at baseline and weeks 12, 24 and 36 by blinded assessment. At FACES, TAU resources for HIV+GBV+ women include medical professionals, counseling, community elders, church leaders, police, and a pro-bono legal aid, all of who have all been involved with past FACES GBV interventions.

ELIGIBILITY:
Inclusion Criteria:

* .(1) HIV+ women enrolled at FACES-Kisumu; (2) Diagnosis with depression (MDD, dysthymia, minor depression) and PTSD secondary to GBV* on the CIDI; (3) Ability to attend weekly therapy sessions and repeated measures; (4) Age greater than 18 years; (5) Ability to give informed consent.

Exclusion Criteria:

* (1) Cognitive dysfunction requiring a higher level of care or compromising ability to participate in IPT**; (2) severe thought or mood disorder symptoms requiring a higher level of care or interfering with ability to participate in IPT; (3) current drug and alcohol dependence requiring substance use treatment. Although PTSD is associated with substance abuse in EuroAmerican populations, a recent study of 5175 FACES patients found that over 80% of this LMIC population use no alcohol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Depression, PTSD | Change from 0-12 weeks, 12-24 weeks and 24-36 weeks
  structured clinical interview: Composite International Diagnostic Interview (CIDI)

SECONDARY OUTCOMES:
ARV adherence | Change from 0-12 weeks, 12-24 weeks and 24-36 weeks
  Visual Analog Scale self-report
HIV viral load | 12 weeks, 24 weeks, 36 weeks
  blood draw

OTHER OUTCOMES:
cost analyses | Cost: 12 weeks; benefits (DALYS and productivity): Change from 0-12 weeks, 12-24 weeks and 24-36 weeks
Neurocognitive outcomes | Change from 0-12 weeks, 12-24 weeks and 24-36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Meffert, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Family AIDS Care Education and Services, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Meffert SM, Neylan TC, McCulloch CE, Blum K, Cohen CR, Bukusi EA, Verdeli H, Markowitz JC, Kahn JG, Bukusi D, Thirumurthy H, Rota G, Rota R, Oketch G, Opiyo E, Ongeri L. Interpersonal psychotherapy delivered by nonspecialists for depression and posttraumatic stress disorder among Kenyan HIV-positive women affected by gender-based violence: Randomized controlled trial. PLoS Med. 2021 Jan 11;18(1):e1003468. doi: 10.1371/journal.pmed.1003468. eCollection 2021 Jan. PMID 33428625
- [Derived] Opiyo E, Ongeri L, Rota G, Verdeli H, Neylan T, Meffert S. Collaborative Interpersonal Psychotherapy for HIV-Positive Women in Kenya: A Case Study From the Mental Health, HIV and Domestic Violence (MIND) Study. J Clin Psychol. 2016 Aug;72(8):779-83. doi: 10.1002/jclp.22359. Epub 2016 Jul 27. PMID 27463639
- [Derived] Onu C, Ongeri L, Bukusi E, Cohen CR, Neylan TC, Oyaro P, Rota G, Otewa F, Delucchi KL, Meffert SM. Interpersonal psychotherapy for depression and posttraumatic stress disorder among HIV-positive women in Kisumu, Kenya: study protocol for a randomized controlled trial. Trials. 2016 Feb 3;17:64. doi: 10.1186/s13063-016-1187-6. PMID 26841875